CLINICAL TRIAL: NCT04710030
Title: Anti Viral Treatment in Mild Cognitive Impairment
Brief Title: Valacyclovir for Mild Cognitive Impairment
Acronym: VALMCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Davangere P. Devanand, Professor of Clinical Psychiatry and Neurology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8089
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment; Herpes Simplex 1; Herpes Simplex 2
Keywords: Valacyclovir; Anti-viral treatment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valacyclovir (Active Comparator): Oral valacyclovir will be distributed in 500mg caplets. Patients will take 8 caplets per day (total dose: 4 grams per day) for 52 weeks.
  Interventions: Drug: Valacyclovir hydrochloride 500mg caplet
- Placebo (Placebo Comparator): The oral placebo (sugar pill) will be distributed in 500mg caplets. Patients will take 8 caplets per day for 52 weeks.
  Interventions: Drug: Placebo sugar pill caplet

INTERVENTIONS:
Drug: Valacyclovir hydrochloride 500mg caplet — Active Comparator
  Other Names: Valtrex
  Arms: Valacyclovir
Drug: Placebo sugar pill caplet — Placebo Comparator
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Anti-viral treatment in Mild Cognitive Impairment (MCI) is a Phase II, placebo-controlled, 52-week trial using oral valacyclovir 4 g/day in 50 HSV seropositive, AD biomarker-positive, amnestic mild cognitive impairment (MCI) patients (eMCI and lMCI). The trial will directly address the long-standing viral etiology hypothesis of Alzheimer's disease (AD) which posits that viruses, particularly the very common herpes simplex virus-1 (HSV1) and herpes simplex virus-2 (HSV2), may be etiologic or contribute to the pathology of AD. This trial will intervene at an earlier stage (MCI). We will compare the repurposed drug valacyclovir to placebo in patients with amnestic MCI (eMCI and lMCI) in a randomized, double-blind, two-arm parallel group 52-week pilot trial. Our Phase II trial will be the first antiviral drug trial conducted in MCI.

DETAILED DESCRIPTION:
Many viruses are latent for decades before being reactivated in the brain by stress, immune compromise, or other factors. After the initial oral infection, herpes simplex virus-1 (HSV1) becomes latent in the trigeminal ganglion and can later enter the brain via retrograde axonal transport, often targeting the temporal lobes.

HSV1 can also enter the brain via olfactory neurons directly. HSV1 (oral herpes) and HSV2 (genital herpes) are known to trigger amyloid aggregation and their DNA is commonly found in amyloid plaques. Anti-HSV drugs reduce Aβ and p-tau accumulation in brains of infected mice. HSV1 reactivation is associated with tau hyperphosphorylation in mice and may play a role in tau propagation across neurons. In humans, recurrent reactivation with newly produced HSV1 particles, 'drop by drop,' may produce neuronal damage and eventually lead to neurodegeneration and Alzheimer's disease (AD) pathology, partly due to effects on amyloid and tau. Clinical studies show cognitive impairment in HSV seropositive patients in different patient groups and in healthy adults, and antiviral treatments show robust efficacy against peripheral HSV infection. The study team will conduct the first-ever clinical trial to directly address the long-standing viral etiology hypothesis of AD which posits that viruses, particularly the very common HSV1 and HSV2, may be etiologic or contribute to the pathology of AD.This trial will intervene at an earlier stage (MCI).

In AD biomarker positive patients with Mild Cognitive Impairment (eMCI and lMCI) who test positive for serum antibodies to HSV1 or HSV2, the generic antiviral drug valacyclovir will be compared at oral doses of 4 grams per day, to matching placebo in the treatment of 50 patients (25 valacyclovir, 25 placebo) in a randomized, double-blind, 52-week Phase II proof of concept trial.

Patients treated with valacyclovir are hypothesized to show smaller decline in cognition and functioning compared to placebo, and, using 18F-Florbetapir PET imaging, to show less amyloid accumulation than placebo over the 52-week trial.

We will explore apolipoprotein E e4 genotype as a moderator, and changes in global clinical status, viral antibodies and proteomic assays, AD signature of MRI regional and whole brain cortical thinning, and plasma total tau, p-tau epitopes and neurofilament light (Nfl) protein markers for neurodegeneration as exploratory hypotheses.

Apolipoprotein biomarker testing will be completed preferably at Week 0 (may be completed at any alternative site visit if necessary), MRI scans at Week 0 and Week 52, PET scans at Screening and Week 52.

This innovative Phase II proof of concept trial clearly has exceptionally high reward potential for the treatment of MCI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 50-95. Females must be postmenopausal, defined as 12 consecutive months without menstruation. (Patient Report)
2. Diagnosis of MCI (includes eMCI and lMCI by ADNI criteria)(Neuropsychological Evaluation)
3. Folstein Mini Mental State (MMSE) greater than or equal to 23/30. (Neuropsychological Evaluation)
4. Patient retains capacity to consent for him/herself. (Physician Evaluation)
5. At screening, patients must test positive for serum antibodies to HSV1 or HSV2. (Laboratory Tests)
6. Use of cholinesterase inhibitors or memantine is not required but will be permitted. If already prescribed, doses of these medications must be stable for 1 month prior to study entry. Patients are permitted to receive cholinesterase inhibitors and/or memantine throughout the duration of the study. Any changes to the medication will be documented in the participant research chart. Medications given for other medical reasons, e.g., antidiabetic or anti-hypertensive medications, will not be altered for the purposes of this trial and the patient's primary physician may adjust such medications as medically indicated throughout the trial. Details of concomitant medication use will be documented at all visits and will be available for statistical analysis.(Patient Report)
7. Either PET amyloid scan positivity at screening, or prior CSF biomarker positive for AD. (Medical Records or through completing a PET scan as part of screening)

Exclusion Criteria:

1. Current clinical diagnosis of schizophrenia, schizoaffective disorder, other psychosis, bipolar disorder or current major depression by DSM-5 criteria. Prior history of major depression will not be exclusionary. (Physician Evaluation)
2. Active suicidal intent or plan based on clinical assessment. (SRMP Assessment by Study Physician)
3. Current or recent (past 6 months) alcohol or substance use disorder (DSM-5 criteria). (Physician Evaluation)
4. Current diagnosis of other major neurological disorders, including Parkinson's disease, multiple sclerosis,CNS infection, Huntington's disease, and amyotrophic lateral sclerosis. (Physician Evaluation)
5. Clinical stroke with residual clinical deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion. (Physician Evaluation)
6. Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases in the last 12 months will be excluded, but past history of successfully treated cancer will not lead to exclusion. (Physician Evaluation)
7. Sitting blood pressure > 160/100 mm Hg. (Physician Evaluation)
8. Renal failure as determined by an estimated Glomerular Filtration Rate (GFR) < 44 ml/min/1.73m2. (Laboratory Report)
9. Serum vitamin B12 levels below the normal range. (Laboratory Report)
10. Patients with thyroid stimulating hormone (TSH) levels above 4.94 mlU/L. (Laboratory Report)
11. Use of benzodiazepines in lorazepam equivalent doses equal to or greater than 2 mg daily. (Patient Report)
12. For MRI, metal implants and pacemaker, and claustrophobia such that the patient refuses MRI. (Patient Report)
13. Radiation exposure in the prior 12 months that, together with 18F- Florbetapir will be above the FDA annual radiation exposure threshold. (Patient Report and Physician Evaluation)
14. Severe vision or hearing impairment that would prevent the participant from performing the psychometric tests accurately. This will be a clinical determination by the study physician without formal testing or audiometry.(Physician Evaluation)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Change in accumulation of amyloid plaque (18F-Florbetapir PET) from Week 0 to Week 52. | Assessed by Week 0 and at Week 52
  18F-Florbetapir PET imaging will show amyloid accumulation in sum of six ROIs (cerebellar gray matter reference) that are known to show increased uptake in AD: medial orbital frontal, anterior cingulate, parietal, temporal, posterior cingulate, precuneus.

SECONDARY OUTCOMES:
Change from week 0 to week 52 in the Alzheimer's Disease Cooperative Study-Preclinical Alzheimer Cognitive Composite (PACC) | Assessed at week 0, week 12, week 26, week 52
  The ADCS-PACC combines four paper-and-pencil cognitive tests: list-learning task from the Free and Cued Selective Reminding Test (FCSRT), paragraph recall test from the Wechsler Memory Scale, Digit Symbol Substitution Test and the Mini-Mental State Examination (MMSE). z-scores are generated from the combination of these test scores. The z-score range is from -5 to +5 with higher scores indicating less deficit and lower scores indicating greater deficit.
Change from week 0 to week 52 in the Alzheimer's Disease Cooperative Study-Activities of Daily Living scale-Prevention Instrument (ADCS-ADL-PI) | Assessed at week 0, week 12, week 26, week 52.
  The ADCS-ADL-PI will be administered to the informant for the assessment of impairments of instrumental and related activities of daily living in patients with MCI. The sum score of the first 15 items in the instrument that indicate impairments in function related to cognition is the outcome. Scores range from 0-45 with lower scores indicating greater functional deficit and higher scores indicating less functional deficit.
Change from week 0 to week 52 in Clinical Dementia Rating (CDR) sum of boxes | Assessed at week 0, week 12, week 26 and week 52.
  The Clinical Dementia Rating is an assessment that evaluates and stages the severity of dementia by scoring a patient's cognitive and functional abilities in six domains. Each domain is rated from 0 (no impairment) to 3 (severe impairment). The total score ranges from 0 to 18 with 0 indicating no impairment and 18 indicating severe impairment.
Change from week 0 to week 52 in Mini Mental Status Exam (MMSE) scores | Assessed at week 0 and week 52.
  MMSE is an assessment of global cognitive performance. Score ranges from 0 to 30 with higher scores indicating better cognitive performance.

OTHER OUTCOMES:
Change from week 0 to week 52 in Magnetic Resonance Imaging (MRI) hippocampal volume | Assessed at week 0 and week 52.
  The average of left and right hippocampal volumes on MRI, determined by using Freesurfer software. Range is 500 to 5,000 cu mm with higher scores indicating larger hippocampal volume
Change from week 0 to week 52 in Magnetic Resonance Imaging (MRI) cortical thickness | Assessed at week 0 and week 52.
  Assessment of thickness of the brain's cerebral cortex, which is the outer layer of gray matter. This is done by using Freesurfer software. The value obtained is by averaging cortical thickness from several brain regions. The range is 0 mm to 5 mm, with higher values indicating greater cortical thickness.
Change from week 0 to week 52 in plasma phosphorylated tau 217 (p-tau217) | Assessed at week 0 and week 52.
  p-tau217 is a blood-based biomarker for Alzheimer's disease that is assayed by the company Quanterix in this study. Values are in pg/ml, range is 0 to 1 pg/ml. Higher values suggest increased likelihood of Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No